CLINICAL TRIAL: NCT00564928
Title: A Phase 2 Open-Label Study to Investigate the Pharmacodynamics and Clinical Activity of IPI-504 in Patients With Castration-Resistant Prostate Cancer Stratified by Prior Chemotherapy
Brief Title: A Phase 2 Study to Investigate the Clinical Activity of IPI-504 in Patients With Hormone-resistant Prostate Cancer
Acronym: IPI-504-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-04
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Cancer of the Prostate
Keywords: Hormone resistant prostate cancer; castrate resistant prostate cancer; HRPC; CRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPI-504: Group A (Experimental): No Prior treatment for prostate cancer with cytotoxic chemotherapy (adjuvant or neoadjuvant chemotherapy is acceptable if completed >2 years prior to study)
  Interventions: Drug: IPI-504
- IPI-504: Group B (Experimental): * Must have evidence of radiographic metastatic disease
  * Must have been treated with a docetaxel-based chemotherapy regimen for HRPC with a minimum of 2 cycles with either PSA or RECIST defined radiographic progression during or witin 60 days of completeing docetaxel based chemotheraph or be intolerant of docetaxel-based chemotherapy
  * No more than three prior chemotherapies regimens for HRPC
  Interventions: Drug: IPI-504

INTERVENTIONS:
Drug: IPI-504 — IPI-504 at 400mg/m2, IV, 2 times a week for 2 weeks with 10 days off treatment. Twenty-one (21) day cycle

SUMMARY:
To determine:

* Anti-tumor activity of IPI-504 in 2 groups of subjects with hormone resistant prostate cancer.
* Group A - subjects who have not previously received chemotherapy
* Group B - sujects who have received prior chemotherapy or could not tolerate chemotherapy.
* Clinical response will be determined by PSA and radiological response

DETAILED DESCRIPTION:
IPI-504 is a novel, water-soluble analog of 17-AAG and a potent inhibitor of Hsp90. Hsp90's role in the cell is to control the proper folding, function, and viability of various "client" proteins. Many of these client proteins (such as AKT, Her-2, Bcr-Abl, PDGFR-α, and c-Kit) are oncoproteins or important cell signaling proteins. Inhibition of HSP-90 leads to the proteasomal degradation of these proteins.

In patients with HRPC,there are several proteins that are important in the progression of HRPC, including AR, AKT and Her-2. All of these are client proteins of Hsp90 and in response to Hsp90 inhibition are degraded by their proteasome. Preclinical studies have shown that Hsp90 inhibition causes a dose dependent degradation of these client proteins and growth inhibition of prostate cancer in xenograft tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Resolution of acute toxic side effects of prior chemotherapy
* Castration resistant disease despite ongoing chemical or surgical castration
* ECOG 0-1
* PSA greater than or equal to 2
* Group A -

  * No Prior treatment for prostate cancer with cytotoxic chemotherapy (neoadjuvant, adjuvant treatment permitted if more than 2 years out)
* Group B

  * Radiographic evidence of metastatic disease
  * Prior tx with docetaxel-minimum of 2 cycles with progression by RECIST or PSA or intolerant of tx
  * Maximum of 3 prior chemotherapies

Exclusion Criteria:

* Small cell carcinoma of the prostate
* Treatment within 2 weeks with approved, investigational, or small molecule
* Treatment within 4 weeks with biologic or external beam radiation
* ANC <1,500 cells m3; Platelets <100,000 mm3; Hemoglobin <9.0g/dL
* AST/ALT >2.5 ULN
* Serum creatinine >3.0mg/dL
* Active keratitis or keratoconjunctivitis
* Previous treatment with 17-AAG, DMAG; or any other HSP-90 inhibitor
* Baseline Qtc >450 mses

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Correlate prior treatment status with clinical response as determined by PSA and radiologic response rate | 12 Weeks

SECONDARY OUTCOMES:
Assess the safety and tolerability of IPI-504 in patients with hormone resistant prostate cancer | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Oh, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - San Bernardino Urological Associates, San Bernardino, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado at Denver, Denver, Colorado
  - MCG Cancer Center, Augusta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Parkland Hospital, Dallas, Texas